CLINICAL TRIAL: NCT03016013
Title: A Phase III Study of RC18,a Recombinant Human B Lymphocyte Stimulating Factor Receptor-Antibody Fusion Protein in Subjects with Poor Efficacy of MTX Due to Treat Moderate and Severe Rheumatoid Arthritis.
Brief Title: A Study of the Efficacy and Safety of TACI-antibody Fusion Protein Injection (RC18) in Subjects with Inadequate Response to MTX Due to Treat Moderate and Severe Rheumatoid Arthritis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C008 RACLLI
Record Dates: First submitted 2017-01-08; First posted 2017-01-10 (Estimated); Last update posted 2024-09-26 (Actual); Status verified 2023-09

CONDITIONS: Moderate and Severe RheumatoId Arthritis
MeSH Terms: conditions — Lymphoma, Follicular; Arthritis, Rheumatoid | interventions — Methotrexate; RC-18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo plus MTX (Placebo Comparator): Patients received placebo SC plus MTX weekly administered subcutaneously for 24 times.All patients had a foundation MTX therapy, MTX dose should be stable, not to adjust the dose. All subjects received RC-18 treatment once a week from week 24 to week 48.
  Interventions: Biological: Placebo plus MTX
- Experimental: RC18 160 mg+MTX (Experimental): Patients received the test group RC18 160mg plus MTX weekly administered subcutaneously for 24 times. All patients had a foundation MTX therapy, MTX dose should be stable, not to adjust the dose.
  Interventions: Biological: RC18 160 mg plus MTX

INTERVENTIONS:
Biological: Placebo plus MTX — The trial was divided into two groups: (1) placebo + MTX; (2) telitacicept 160 mg + MTX. MTX was used as the basic treatment, the dose of MTX was stable during the trial, and could not be adjusted. Telitacicept or placebo was administered once a week for the first 24 weeks. Beginning at week 24, subjects in the placebo group will enter the RC-18 treatment group. All subjects received RC-18 treatment once a week from week 24 to week 48.
  Other Names: MTX=Methotrexate
  Arms: Placebo plus MTX
Biological: RC18 160 mg plus MTX — The trial was divided into two groups: (1) placebo + MTX; (2) telitacicept 160 mg + MTX. MTX was used as the basic treatment, the dose of MTX was stable during the trial, and could not be adjusted. Telitacicept or placebo was administered once a week for the first 24 weeks. Beginning at week 24, subjects in the placebo group will enter the RC-18 treatment group. All subjects received RC-18 treatment once a week from week 24 to week 48.
  Other Names: RC18; MTX=Methotrexate
  Arms: Experimental: RC18 160 mg+MTX

SUMMARY:
The purpose of this study is to initially access the safety and effectivity of RC18 combined with methotrexate (MTX) in comparison with the use of methotrexate alone in participants with moderate to severe Rheumatoid Arthritis (RA) who have an inadequate response to MTX therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult onset RA by a physician as defined by the 1987 and/or 2010 ACR criteria and ESR or C - reaction protein ( CRP ) is greater than the normal range;
* Aged 18-65 years old;
* Consent to use effective contraception during the study period (women of childbearing age);
* Patients with an inadequate response to existing therapies at least one anti-TNFs Infliximab (Remicade ) at least three times, adalimumab (Humira), at least four times, etanercept ( Enbrel) use at least 8 weeks, etanercept use at least 8 weeks.And Last medication time to randomization more than 12 weeks;
* Voluntarily signed informed consent;
* Patients have been taking MTX for at least 12 weeks at the screening and maintaining dose stability ≥7.5mg/ weeks (or equivalent dose) 4 weeks before randomization;
* Treatment with traditional oral disease-modifying antirheumatic drugs (DMARD) /immunosuppressive agents other than MTX within 4 weeks or 12 weeks before the screening visit, depending on DMARD;
* If subjects are receiving treatment of corticosteroid, must stabilize dose (dose of prednisone) at least equal to or less than 10mg/day for 4 weeks (before randomization);
* If subjects are receiving treatment of NSAIDs,must stabilize dose (dose of prednisone) at least 4 weeks (before randomization);
* When the patient's condition to achieve moderate to severe active RA at the screening, defined as at least 6/68 tenderness joints and at least 6/66 swollen joints.

Exclusion Criteria:

* Exclusion criteria associated with rheumatoid disease:

  1. The subjects with any other inflammatory arthritis (such as juvenile chronic arthritis, regional enteritis (Krohn S disease), ulcerative colitis, gout, active vasculitis, psoriatic arthritis or ankylosing spondylitis);
  2. The subjects with secondary, non inflammatory arthritis (such as osteoarthritis or fibromyalgia), and researchers think the symptoms of arthritis can interfere with judgment and evaluation study on therapeutic effects of drugs.But secondary Sjogren syndrome (SjÖgren), thyroiditis without exclusion;
  3. The subjects had a history of prosthetic joint infection, whenever the infection occurred, and the artificial joint is still in the body;
  4. The subjects due to RA and/or shoulder hand syndrome IV grade received more than 3 times the arthroplasty;
  5. The subjects' Types of X-ray phases reach IV phase.
* The subjects can not accept the prohibited drugs listed in the following table:

  1. Use of analgesics (acetaminophen / paracetamol) within 24 hours before baseline assessment;
  2. dosage regimen of nonsteroidal anti-inflammatory analgesic NSAIDs/COX-2 inhibitors (except acetaminophen) have occurred any change within 14 days before baseline assessment;
  3. The dosage of oral glucocorticoids have occurred any change within 28 days before baseline assessment;
  4. Intramuscular injection/intravenous injection/intra-articular injection of glucocorticoid has used within 28 days before baseline assessment;
  5. Intra-articular injection of hyaluronic acid has used within 28 days before baseline assessment;
  6. Tripterygium wilfordii or other traditional Chinese medicine for treating RA has used within 28 days before baseline assessment.
* The researchers confirmed that the subjects had current or recent severe, progressive and or not controlled heart, lung, liver, kidney and other important organs and blood, endocrine system lesions and history; Abnormal laboratory parameters need to be excluded, including but not limited to:

  1. Cr >135μmol/L or 5 times the upper limit of laboratory reference value;
  2. WBCs<3x 109/L;
  3. neutrophile granulocyte <1.5×109/L;
  4. hemoglobin<85g/L;
  5. platelet count<80x 109/L;
  6. total bilirubin > 1.5 times the upper limit of laboratory reference value;
  7. AST > 2 times the upper limit of laboratory reference value;
  8. ALT > 2 times the upper limit of laboratory reference value;
  9. alkaline phosphatase > 2 times the upper limit of laboratory reference value.
* HBsAg-surface antigen positive patients are not allowed to be selected, but only anti HBC single positive is added to do HBV-DNA quantitative detection, if the HBV-DNA quantity is negative can not be regarded as the exclusion.
* The anti-HCV of patients show positive.
* Infection with herpes zoster or HIV virus at the screening.
* The subjects at high risk of infection ;such as leg ulcers, indwelling catheter, persistent or recurrent chest infection, completely bedridden or sedentary wheelchair subjects.
* There is a history of chronic infection, severe or life-threatening infections (including shingles) within the last 6 months, or any signs or symptoms during the screening period that may indicate an infection (e.g. fever, cough).
* the subjects currently or recently (30 days before screening) suffers from severe viral, bacterial, fungal, or parasitic infections.
* pregnant, lactating women and men or women who have birth plans in the past 6 months.
* Have a history of allergic reaction to contrast agent for parenteral administration and human biological medicines.
* The subjects receive live vaccine/attenuated vaccine within the first 8 weeks before screening or those who are known to receive live vaccine/attenuated vaccine during the trial.
* Have participated in any clinical trial in the first 28 days of the initial screening or 5 times half-life period of the study compound (taking the time for the elderly).
* Patients with using of biological agents for the treatment of DMARDs within three months.
* Active TB at screening.Exception for patients with PPD≥15mm.But Patients with anti tuberculosis treatment for 3 years without relapse are allowed to participate in the trial.
* Malignant tumor patients :the patients who suffering from malignant tumor has been removed and no recurrence or who with cervical carcinoma in situ have evidence of metastatic disease and with basal cell or squamous cell carcinoma had been completely removed and at least 3 years without recurrence can participate in.
* The patients with a history of lymphoproliferative disease (including lymphoma or signs and symptoms of lymphoproliferative disease at any time).
* the patients have no effective in using of tumor necrosis factor inhibitors;
* there was a history of long-term alcohol abuse, intravenous drug abuse or other illicit drug abuse within 6 months.
* Planning to have surgery for RA or other significant surgery during the period of the study.
* patients experienced any of the following events within 12 weeks before screening: myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association class IV heart failure.
* Patients received interferon treatment (such as interferon alpha, intron alpha, peg-intron, double talon, intergen, Pegasys etc.) within 4 weeks before screening,or are expected to test period will need to accept interferon therapy.
* The combined use of immunosuppressive agents associated with organ. transplantation is not allowed during the study period.
* Immunosuppressive agents associated with organ transplantation should not be allowed during the study period.
* Investigator considers candidates not appropriating for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in each group reached ACR20 at week 24 | Week 24（Visit 9）
  ACR20 response: Patients with tenderness and swollen joint counts and 20% improvement,At least 3 20% improvement in the following 5:a.Health Assessment Questionnaire;b.Subjects assessed pain VAS score;c.Assess the overall situation of the disease subject VAS score;d.Researchers assessed the overall situation of the disease in the VAS score;e.Acute phase reactants(ESR or CRP).

SECONDARY OUTCOMES:
Percentage of Participants Achieving American College of Rheumatology ACR50 and ACR70 Responses at week 24. | Week 24
Percentage of Participants Achieving Low Disease Activity and clinical remission. (DAS28 ≤3.20 and DAS28 < 2.6). | Week 24
  Disease activity score based on 28 painful joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR) mm/hr, and general health (GH) using a visual analog scale (VAS); VAS range: 0 (very well) to 100 (extremely bad). DAS28 score calculated as 0.56 √ (28 painful joint count) + 0.28 √ (28 swollen joint count) + 0.70 (ln ESR mm/hr) + 0.014 GH; range 0 to 10. DAS28 score >5.10=higher disease activity; <3.20=low disease activity; <2.60=clinical remission.
Percentage of Participants Achieving American College of Rheumatology ACR50 and ACR70 Responses at week 12 or week 24. | Week 12 and Week 24
Sharp Score Relative Change from Baseline at Week 24 | Week 24
Percentage of Participants With American College of Rheumatology 20% ,50% and 70% (ACR20, ACR50 and ACR70) Response | Week 4, Week 8, Week 12, Week 28, Week 32, Week 40, Week48
Change From Baseline in Joint Space Narrowing and Erosions at week 24 and week 48. | Week 24,Week48
  Erosion score (a component of the modified TSS) is a measure of change in joint health. Erosion score range is from 0 (no erosion) to 280 (high erosion).And Joint space narrowing score (a component of the modified TSS) also is a measure of change in joint health. Joint space narrowing score range is 0 (no narrowing) to 168 (high narrowing).

CONTACTS AND LOCATIONS:
Overall Officials: Fengchun Zhang, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided